CLINICAL TRIAL: NCT04483141
Title: Translation and Validation of the Abbey Pain Scale in Stroke Patients
Brief Title: Translation and Validation of the Abbey Pain Scale in Stroke Patients (ABBEY-F)
Acronym: ABBEY-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 FERRIER; 2020-A01360-39 (Other: ANSM)
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Pain
Keywords: stroke; pain; aphasia; Abbey pain scale
MeSH Terms: conditions — Stroke; Pain; Aphasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-communicant stroke patients: Patients suffering from stroke, and unable to efficient communication. They will be assessed for pain through several tools (hetero-assessment of pain).
  Interventions: Diagnostic Test: Abbey Pain Scale
- communicant stroke patients: Patients suffering from stroke, and unable to efficient communication. They will be assessed for pain through several tools (including hetero-assessment and auto-assessment of pain)
  Interventions: Diagnostic Test: Abbey Pain Scale

INTERVENTIONS:
Diagnostic Test: Abbey Pain Scale — Hetero-assessment of pain

SUMMARY:
Pain is common after a stroke, affecting up to 49% of patients within 2 years of the event. They include headache, musculoskeletal pain, spasticity and central neuropathic pain. A wide range of patients have communication problems after stroke that make it difficult to assess pain. Yet there is a major impact of pain on the quality of life of these patients. Some tools have been validated to assess pain in non-communicative patients, but none are specific to stroke patients. The Algoplus scale is commonly used in intra-hospital care in France. The Abbey Pain Scale is not translated into French, and could provide a more accurate pain rating for non-communicative patients.

The objective is to validate a French version of the Abbey Pain Scale for stroke patients.

It is an observational study with longitudinal data collection. It is planned to include 120 patients from the neurology department of the Clermont-Ferrand University Hospital.

DETAILED DESCRIPTION:
The study will be conducted over a 12-month period. 120 patients hospitalized for stroke including 60 communicating and 60 non-communicating patients will be recruited. Epidemiological data will be collected at enrollment, as well as an initial assessment using the Abbey and Algoplus scales for non-communicating and communicating patients, and also the numerical scale for communicating patients. The HADS questionnaire will be completed by communicating patients only. Of the 60 patients in each group, 30 will receive a second concurrent assessment by an inter-rater, 30 will receive a test/retest reassessment after 30 minutes, and 20 will be reassessed 90 minutes later by the same scales after pain treatment. For 30 of the 120 patients, an infrared pupillometry measurement will be performed before and after treatment of acute pain. All patients will be recruited from the neurovascular unit of the Clermont-Ferrand University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old ;
* Covered by Social Security;
* Hospitalized in the Neurovascular Unit for the management of ischemic stroke with or without reperfusion treatment, or hemorrhagic stroke;
* NIHSS score greater than 1;
* For communicating patients: French mother tongue, or reading French without assistance, and able to understand the objectives.

Exclusion Criteria:

* Refusal ;
* Legally protected patient
* Pregnancy;
* Pre-stroke psychiatric or neurodevelopmental disorders;
* Transient ischemic attack;
* Specific strokes: Bithalamic, locked-in syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in the Neurovascular Unit for the management of ischemic stroke with or without reperfusion treatment, or hemorrhagic stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Abbey Pain Hetero-Evaluation Scale | day 0
  This scale searches for elements suggestive of pain in the patient by scoring between 0 (absent) and 3 (severe) each of the items: vocalization, facial expression, body language, physiological modifications, physical modifications; obtaining a score between 0 and 18.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale (HADS) Questionnaire | day 0
  This scale is an instrument to screen for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions relate to the anxiety dimension (total A) and seven others to the depressive dimension (total D), giving 2 scores. for communicant patients only
Algoplus Pain Hetero-Evaluation Scale | day 0
  This scale searches for elements suggestive of pain in the patient by answering YES/NO to each of the items: face, gaze, complaints, body, and behaviour; score between 0 and 5.
Numerical Scale | day 0
  This is a communicant patient's self-assessment of the intensity of pain felt, between 0 (no pain) and 10 (maximum pain). for communicant patients only
Infrared pupillometry measurement | day 0 before treatment of acute pain
  It is an absolute measurement of pupil size using a portable pupillometer
Infrared pupillometry measurement | day 0 after treatment of acute pain
  It is an absolute measurement of pupil size using a portable pupillometer

CONTACTS AND LOCATIONS:
Overall Officials: Anna FERRIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France